**Unique Protocol ID: No.2023023** 

Official Title: Effects of transcranial direct current stimulation combined with retrieval practice on semantic memory in patients with schizophrenia

**Document Title: Informed Consent** 

Date of the Document: 2024/7/31

## **Informed Consent**

| Clinical Research | Program | : Effec | ets of tran | iscrai | nial direct | current st | imul | ation com | bined |
|---|---|---|---|---|---|---|---|---|---|
| | with r | etrieval | practice | on | semantic | memory | in | patients | with |
| | schizop | hrenia | _ | | | _ | | | |
| Project Organizer: | | Northwest Normal University | | | | | | | |
| Project Collaborate | ors: | Th | e Third Pe | ople' | s Hospital o | of Lanzhou | 1 | | |

## **Statement of Consent**

Dear Patient:

We would like to invite you to participate in a study on the effects of extraction exercises combined with transcranial direct current stimulation on memory in patients with schizophrenia. The study protocol has been reviewed and approved by the Ethics Committee of Northwest Normal University and the Third People's Hospital of Lanzhou City for clinical research.

I am aware of the possible risks and benefits of participating in this study. The experimenter has answered all questions about this study. I confirm that I have had sufficient time to participate in this study and agree to the following:

- I am volunteering to participate in this study.
- I may ask my doctor for more information at any time.
- I can withdraw from this study at any time without discrimination or retaliation, and my medical treatment and rights will not be affected.

Finally, I have decided to agree to participate in this study and promise to follow my doctor's instructions as much as possible.

## Patient's signature:

I confirm that the details of this trial have been explained to the patient, including its powers and possible benefits and risks.

Signature of the doctor: